CLINICAL TRIAL: NCT06159959
Title: Carbetocin in the Prevention of Primary Postpartum Haemorrhage in Obese Versus Non-obese Women Undergoing Elective Cesarean Section
Brief Title: Carbetocin in the Prevention of Primary Postpartum Haemorrhage
Status: Completed | Type: Observational
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, Dina Sanad Tawfik Allam, Specialist of Obstetrics and Gynecology at AlSahelTeaching Hospital, Ministry of Health and Population, Egypt
Other Study IDs: Dina Sanad Tawfik
Record Dates: First submitted 2023-11-25; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Post Partum Hemorrhage
Keywords: Obesity; PPH; BMI; Carbetocin; Oxytocin; Uterotonic
MeSH Terms: conditions — Postpartum Hemorrhage; Obesity | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Obese Pregnant Females: About 122 Pregnant women candidate for elective cesarean section suffering from obesity where as Body mass index (BMI) is ≥30 kg/m2
  Interventions: Drug: Carbetocin
- Group B: Non-Obese Pregnant Females: About 122 Pregnant women candidate for elective cesarean section and not obese obesity where as Body mass index (BMI) is < 30 kg/m2
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — To assess the effectiveness of single IV bolus dose of carbetocin in the prevention of primary PPH in obese versus non obese women undergoing elective cesarean section.
  Other Names: Oxytocin

SUMMARY:
Postpartum haemorrhage (PPH) ranks as the first cause of maternal mortality in developing countries and it is the cause of 25% of maternal deaths worldwide.

Carbetocin is a long-acting synthetic octapeptide analogue of oxytocin with agonist properties. Like oxytocin, carbetocin binds to oxytocin receptors present on the smooth musculature of the uterus, resulting in rhythmic contractions of the uterus, increased frequency of existing contractions and increased uterine tone.

DETAILED DESCRIPTION:
Postpartum hemorrhage is defined as a blood loss more than 500 ml, and serious PPH as a blood loss more than 1,000 ml.

It is a common maternal morbidity in high-resource countries and is trending upward and prevention of postpartum haemorrhage is, therefore, of great importance for improved maternal health care.

Although two-thirds of the PPH cases occur in women without predisposing factors, there are several risk factors for PPH. The most frequent cause of PPH is uterine atony, contributing up to 80 % of the PPH cases .

Studies investigating effect of increased BMI on birth outcomes in a general obstetric population revealed an association between obesity and PPH. The overall increased risk of postpartum hemorrhage among obese women was 8-13%, depending on obesity class.

The risk of postpartum haemorrhage is much higher for women undergoing Cesarean section, particularly in developing countries, where the majority of operations are carried out as an emergency procedure.

Maternal obesity is associated with an elevated risk of intrapartum cesarean section, mainly due to reduced uterine contractility culminating in failure to progress in labor .

Up to date, which uterotonic agent suitable for prophylactic use is being debated and literature lacks of clear endpoints on this item .

The most routinely and widely used uterotonic agent for preventing postpartum haemorrhage is oxytocin, but it only has a half-life of 4-10 min. So, it must be administered as a continuous intravenous infusion to achieve sustained uterotonic activity, which is inconvenient and makes dosing errors a possibility.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40years.
* Body mass index (BMI): Obese ≥30 kg/m2 and non-obese women <30 kg/m2 calculated using maternal height and weight measured to the nearest centimeter and kilogram, respectively, at time of admission to labor word.
* Gestational age: Gestational age ≥37 weeks (gestational age will be recorded according to the last menstrual period and confirmed by ultrasound). In case of discrepancy, a 1st trimesteric ultrasound will be taken as the actual gestational age.
* Singleton pregnancy.

Exclusion Criteria:

Patients who have any factors that might increase the risk of postpartum haemorrhage will be excluded as anemic patients (Hb<10.5g%), antepartum haemorrhage ( placenta previa, placental abruption ), uterine myomata, multiple gestation, polyhydramnios.

* Patients with pre-existing bleeding or thromboembolic disorder.
* Patients with chronic medical diseases (cardiac, hepatic, renal)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: To assess the effectiveness of single IV bolus dose of carbetocin in the prevention of primary PPH in obese versus non obese women undergoing elective cesarean section.
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Post postpartum bleeding | first 6 hours after the Cesarean Section
  To compare the incidence of primary postpartum hemorrhage in both groups receiving carbetocin

SECONDARY OUTCOMES:
Sever PPH as bleeding is >1000 cc | first 24 hours after Cesarean Section
  Outcome of the study will be measured in terms of assessment of Hemoglobin level and Hematocrit level post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Y Elkateb, Professor, Study Chair — Cairo University
Locations (1):
- Kasr- Alainy Hospitals, Cairo, Egypt